CLINICAL TRIAL: NCT01180582
Title: Prospective Clinical Study Using Roentgen Stereophotogrammetric Analysis (RSA) and DEXA to Evaluate Fixation of Periapatite Coated Triathlon Total Knee Arthroplasty Components
Brief Title: Roentgen Stereophotogrammetric Analysis (RSA) and Dual Energy X-ray Absorptiometry (DEXA) to Evaluate Fixation of Periapatite Coated Triathlon Total Knee Arthroplasty (TKA) Components
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Stryker Orthopaedics (Industry); Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Michael Dunbar, MD, PhD, Dalhousie University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDHA-RS/2009-039
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Osteoarthritis, Knee
Keywords: knee; arthroplasty; RSA; migration; micromotion; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Triathlon Periapatite (PA)-coated Tibial Component — Triathlon Periapatite (PA)-coated Total Knee Arthroplasty Tibial Component for uncemented fixation

SUMMARY:
The purpose of this study is twofold: 1) to use RSA to determine the migration patterns of the PA coated Triathlon Total Knee Arthroplasty components during the first 2 years postoperatively and thus determine the proportion of cases where adequate fixation is achieved, and 2) to use DEXA scanning to document peri-prosthetic bone mineral density changes in response to the PA coated Triathlon Total Knee arthroplasty over the first two postoperative years.

In addition, gait assessment and validated outcome questionnaires will be utilized to quantify changes in functional status of subjects after surgery and migration patterns will be compared to results obtained from previous studies of uncemented total knee arthroplasty components conducted at this centre. Questions to be asked are: 1. Do the components achieve adequate fixation to the underlying bone? 2. What are the migration patterns (translations and rotations) of the PA coated arthroplasty components during the first two years postoperatively and are they different from that seen for other implants that have been studied with RSA at this institution? 3. For what proportion of implants does migration continue to increase during the two year follow-up? 4. Are inducible displacements, measured at weight-bearing follow-ups, consistent over time and do they indicate that adequate fixation has been achieved? 5. Are there changes over time in bone mineral density of peri-prosthetic bone in the PA coated Triathlon total knee arthroplasty? 6: Where do changes in bone mineral density occur? 7: Is there a significant difference in health status and functional outcome before and after total knee arthroplasty using PA coated Triathlon total knee arthroplasty components? 8: Are there changes in gait symmetry and centre of mass (COM) displacements as assessed with the Walkabout Portable Gait Monitor pre- and post-operatively and how does study gait data compare to asymptomatic gait? and finally, Question 9: Are there differences in the micromotion patterns between the when compared to other samples of knee implants in our RSA database?

ELIGIBILITY:
Inclusion Criteria:

* symptomatic osteoarthritis of the knee indicating surgical intervention
* ability to give informed consent

Exclusion Criteria:

* significant co-morbidity affecting ability to ambulate
* range of motion measurements that are beyond the realm of normal
* a BMI > 40 (morbid obesity)
* severe osteoporosis or osteopenia or neuromuscular impairment
* women who are pregnant will also be excluded due to the risks of the surgery

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Migration of tibial component as measured with RSA | 2 years

SECONDARY OUTCOMES:
Bone mineral density | 2 years
Subjective health outcome questionnaires - SF-36, WOMAC, Knee Society Function Score, Pain Catastrophizing Scale (PCS), Self-Administered Comorbidity Questionnaire (SCQ) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Dunbar, FRCSC, PhD, Principal Investigator — Dalhousie University & Capital District Health Authority
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada